CLINICAL TRIAL: NCT00770744
Title: A Randomised, Double-blind, Parallel-group, Active-controlled, Flexible Dose Study Exploring the Efficacy and Safety of 12 Weeks Treatment With Lu 31-130 in Patients With Schizophrenia
Brief Title: Efficacy of Lu 31-130 in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12396A; 2008-000479-11 (EudraCT Number)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic; Olanzapine; Lu 31-130
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zicronapine (Experimental)
  Interventions: Drug: Zicronapine
- Olanzapine (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Zicronapine — 5-7mg/day; orally, encapsulated tablets, once daily
  Other Names: Lu 31-130
  Arms: Zicronapine
Drug: Olanzapine — 10-15mg/day; orally, encapsulated tablets, once daily
  Other Names: Zyprexa
  Arms: Olanzapine

SUMMARY:
The main purpose with the study is to explore the efficacy and safety of Lu 31-130 in patients suffering from schizophrenia compared to a standard antipsychotic drug.

DETAILED DESCRIPTION:
Schizophrenia is a serious and disabling mental disorder that affects approximately 1% of the world's population. Antipsychotic drugs remain the cornerstone in the pharmacotherapy of schizophrenia. However, none of the available drugs is ideal, in particular because of their complex safety profile and the limited effectiveness against certain symptom domains. Whereas positive symptoms respond to treatment the effects on negative symptoms and cognitive impairment are only very modest.

Thus present treatment options leave room for improvement and call for new, more effective pharmacotherapies for the treatment of schizophrenia. In the current study, patients suffering from schizophrenia and experiencing clinically significant symptoms of the disease will be included. Eligible patients will be randomised to blinded treatment with either flexible doses of Lu 31-130 or flexible doses of a standard antipsychotic treatment (olanzapine) for 12 weeks. The efficacy (including potential effects on cognitive symptoms) and the safety of Lu 31-130 will be explored in comparison to olanzapine.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a primary diagnosis of schizophrenia
* The subject experiences clinically significant symptoms
* The subject is willing to be hospitalized during the initial period of the study
* The subject has normal serum values of parameters associated with liver function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-09; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change in the Positive and Negative Syndrome Scale (PANSS) score from Baseline to Week 12 | 12 weeks

SECONDARY OUTCOMES:
Change in cognitive symptoms using Assessment of Cognition in Schizophrenia (BACS) test battery. Change in Clinical Global Impression/Improvement (CGI-S/I) scores. Change in Calgary Depression Scale for Schizophrenia (CDSS) score. Safety assessments. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (21):
- Czechia (6):
  - CZ001, České Budějovice
  - CZ005, Litoměřice
  - CZ004, Lnáře
  - CZ002, Olomouc
  - CZ003, Olomouc
  - CZ006, Prague
- France (3):
  - FR001, Clermont-Ferrand
  - FR002, Dole
  - FR003, Jonzac
- HK001, Hong Kong, Hong Kong
- Indonesia (2):
  - ID001, Bangli
  - ID002, Jakarta
- Philippines (2):
  - PH002, Baguio City
  - PH001, Mandaluyong
- Poland (2):
  - PL003, Gdansk
  - PL002, Lodz
- Spain (3):
  - ES001, Barcelona
  - ES002, Salamanca
  - ES004, Zamora
- Thailand (2):
  - TH001, Bangkok
  - TH002, Chiang Mai

REFERENCES:
- Available data/document: EMA EudraCT Results: 2008-000479-11 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2008-000479-11/results